CLINICAL TRIAL: NCT00697580
Title: Intra-Abdominal Fat and Risk of Disease in Adolescents
Brief Title: Strength and Nutrition Outcomes for Latino Adolescents
Acronym: SANO LA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michael I. Goran, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD033064 (NIH); 5R01HD033064 (NIH)
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Type 2 Diabetes; Cardiovascular Risk; Cancer
Keywords: Obesity; Type 2 Diabetes; Cardiovascular risk; Cancer; Latino; Adolescents; Strength Training; Circuit Training; Nutrition
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Neoplasms | interventions — Nutritional Status; Resistance Training; Circuit-Based Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): Control (C)
- 2 (Experimental): Nutrition (N)
  Interventions: Behavioral: Nutrition
- 3 (Experimental): Strength Training & Nutrition (ST + N)
  Interventions: Behavioral: Strength Training & Nutrition
- 4 (Experimental): Circuit Training & Nutrition (CT + N)
  Interventions: Behavioral: Circuit Training & Nutrition

INTERVENTIONS:
Behavioral: Nutrition — Nutrition classes for 1 hour & 30 minutes once a week for 16 weeks + motivational interviewing (4 individual sessions)
  Arms: 2
Behavioral: Strength Training & Nutrition — Strength Training twice a week for 1 hour a day for 16 weeks + Nutrition once a week for 1 hour & 30 minutes for 16 weeks + motivational interviewing (4 individual & 4 group sessions)
  Arms: 3
Behavioral: Circuit Training & Nutrition — Circuit Training twice a week for 1 hour a day for 16 weeks + Nutrition once a week for 1 hour & 30 minutes for 16 weeks + motivational interviewing (4 individual & 4 group sessions)
  Arms: 4

SUMMARY:
We are conducting an intervention study to examine the effects of a 16-week exercise and diet interventions on prevention of disease, specifically type 2 diabetes and heart disease, in Latino youth. Eighty overweight Latino boys and girls will be recruited and placed in one of the following intervention groups: 1) Control Group (delayed intervention), 2) Dietary Education Group (nutrition education focused on reducing sugar & soda, increased fiber & whole grain intake), 3) Combination of Strength Training (twice/week for 60 min, progressive increases in exercise volume and intensity) + Dietary Education (nutrition education focused on reducing sugar & soda, increased fiber & whole grain intake) or 4) Combination of Circuit Training (twice/week for 60 min, aerobic + strength training exercises) + Dietary Education (same as above). We will assess which intervention group has the most effects on health parameters such as weight, body composition, and insulin related measures.

DETAILED DESCRIPTION:
The overall historical goal of this grant has been to examine the determinants of insulin resistance in children, especially the role of total fat and visceral fat during pubertal development in "high risk" minority children. Our previous longitudinal work has provided the platform to propose a new intervention phase of this research. This new emphasis is justified based on the magnitude of the pediatric obesity problem, particularly in susceptible ethnic groups, and the need to design and test novel interventions to reduce not just obesity, but the profound insulin resistance that we have observed in overweight minority children. Insulin resistance is thought to be central (and perhaps causative) to several metabolic abnormalities associated with type 2 diabetes and cardiovascular disease. Thus, interventions aimed at improving insulin resistance in susceptible children could be an effective means in the primary prevention of type 2 diabetes and cardiovascular disease.

The overall objective of this proposal is therefore to conduct a randomized controlled study to examine the effects of 16-week exercise and diet interventions on insulin sensitivity, insulin secretion, beta-cell function, and body fat distribution. Overweight Hispanic boys and girls (n=80) will be recruited and randomized to one of the following interventions:

Ø Control (delayed intervention) Ø Modification of carbohydrate intake (reduced sugar & soda, increased fiber & whole grain intake) using an individualized healthy exchange system and motivational interviewing Ø Strength training + modification of carbohydrate intake Ø Circuit Training + modification of carbohydrate intake

This study will provide new information on the effects of these interventions on primary outcomes at the level of body composition (total lean and fat mass, visceral fat, intramyocellular fat and liver fat) and insulin related measures (insulin secretion & sensitivity and beta-cell function). The hypotheses are:

1. All interventions will have separate and independent effects on improving insulin resistance
2. Strength training will improve insulin resistance by re-distribution of body fat (lower visceral fat, intramyocellular lipid and liver fat)
3. Carbohydrate modification will improve insulin secretion and beta-cell function
4. Circuit training will have similar improvements in insulin resistance and have more improvements on adiposity compared to the strength training group.
5. The aforementioned effects on insulin dynamics will be independent of any effects of either intervention on weight loss or loss in whole body fat.

The overall rationale for these interventions is based on three main factors. First, preliminary data are presented in overweight Hispanic boys showing that 16-weeks of strength training significantly improves insulin sensitivity in the absence of a reduction in total body fat and in the absence of any dietary intervention. Second, preliminary data suggests that overweight Hispanic children consume high levels of simple sugar, and low levels of fiber and complex carbohydrates, and data from the literature suggests that modification of carbohydrate consumption (reduced sugar, increased fiber & whole grain) can improve glucose control independent of body composition. Third we provide new preliminary data showing that the only dietary variable associated with insulin dynamics in overweight Hispanic children was high sugar intake which was associated with poor beta-cell function.

We have chosen to focus on Hispanic children because they are an understudied, high-risk population, and display significant obesity-related metabolic abnormalities probably emanating from profound insulin resistance (see preliminary data). In support of the feasibility of our proposal, we have developed extensive expertise in recruiting and retaining research volunteers from the large Hispanic population of East Los Angeles, we have an experienced multi-disciplinary group of investigators, and the University of Southern California has the necessary clinical research infrastructure to tackle this project. If our hypotheses are borne out, it will provide evidence for the incorporation of strength training and more specific and individualized dietary recommendations in the prevention and management of obesity, type 2 diabetes, and cardiovascular risk in overweight Hispanic youth.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (age- & sex-specific body mass index ≥ 85th percentile based on CDC BMI growth charts [US Department of Health and Human Services, 2000], calculated by Epi Info Software, version 3.3)
* Latino (both sets of grandparents must be of Latino heritage as defined by self-report; limited to Latinos to maintain a homogeneous sample and because Latinos are at increased risk of insulin resistance and type 2 diabetes.) If the participant or the parent is unsure of the country of origin of all 4 grandparents they will be excluded from the study. The participants and their families are not asked whether or not their grandparents are undocumented immigrants.

Exclusion Criteria:

* Presently taking medication(s) or diagnosed with any syndrome or disease that could influence dietary intake, exercise ability, body composition and fat distribution, or insulin action and secretion.
* Previously diagnosed with any major illness since birth (e.g. severe intrauterine growth retardation, chronic birth asphyxia, cancer).
* Children will not be eligible for participation if they have any diagnostic criteria for diabetes including polyuria, polydipsia with or without unexplained weight loss, fasting plasma glucose > 126 mg/dl, or a 2-hour plasma glucose >200 mg/dL during an oral glucose tolerance test. Children will also be excluded if they test positive for diabetes-related auto-antibodies, including ICA512 and GAD. Children testing positive for type 2 diabetes will be referred for treatment. Children with impaired glucose tolerance (fasting glucose >110 mg/dL or 2-hour glucose >140 mg/dl during an OGTT) and/or conditions associated with insulin resistance (e.g. acanthosis nigricans, hypertension, dyslipidemia, PCOS) will be eligible, as long as they are not receiving treatment and meet other eligibility criteria.
* Participants who are involved in any weight training, exercise, nutrition, or weight loss program or have been in the past 6 months.
* Participants that do not follow the rules and guidelines of appropriate conduct during participation, i.e., disruptive behavior, derogatory or racist comments, or any acts of physical violence towards study staff or other participants, and use of illegal substances. The principal investigator Dr. Michael Goran will decide if this conduct warrants exclusion or removal from the study.
* Pregnancy test comes out positive.
* Children who live further than 20 miles away from the General Clinic Research Center (GCRC).
* We can terminate participation if the child fails to follow the rules and guidelines of appropriate behavior and conduct during participation.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2005-05; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | post intervention (week 16)

SECONDARY OUTCOMES:
adiposity | post-intervention (week 16)

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, PhD, Principal Investigator — University of Southern California
Locations (1):
- Veronica Atkins Lifestyle Intervention Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gyllenhammer LE, Alderete TL, Mahurka S, Allayee H, Goran MI. Adipose tissue 11betaHSD1 gene expression, betacell function and ectopic fat in obese African Americans versus Hispanics. Obesity (Silver Spring). 2014 Jan;22(1):14-8. doi: 10.1002/oby.20571. Epub 2013 Sep 10. PMID 23836520
- [Derived] Hasson RE, Adam TC, Davis JN, Watanabe RM, Goran MI. Compensatory responses to insulin resistance in obese African-American and Latina girls. Pediatr Obes. 2013 Dec;8(6):e68-73. doi: 10.1111/j.2047-6310.2013.00184.x. Epub 2013 Jul 2. PMID 23818490
- [Derived] Le KA, Mahurkar S, Alderete TL, Hasson RE, Adam TC, Kim JS, Beale E, Xie C, Greenberg AS, Allayee H, Goran MI. Subcutaneous adipose tissue macrophage infiltration is associated with hepatic and visceral fat deposition, hyperinsulinemia, and stimulation of NF-kappaB stress pathway. Diabetes. 2011 Nov;60(11):2802-9. doi: 10.2337/db10-1263. PMID 22025778
- [Derived] Le KA, Ventura EE, Fisher JQ, Davis JN, Weigensberg MJ, Punyanitya M, Hu HH, Nayak KS, Goran MI. Ethnic differences in pancreatic fat accumulation and its relationship with other fat depots and inflammatory markers. Diabetes Care. 2011 Feb;34(2):485-90. doi: 10.2337/dc10-0760. PMID 21270204
- [Derived] Davis JN, Le KA, Walker RW, Vikman S, Spruijt-Metz D, Weigensberg MJ, Allayee H, Goran MI. Increased hepatic fat in overweight Hispanic youth influenced by interaction between genetic variation in PNPLA3 and high dietary carbohydrate and sugar consumption. Am J Clin Nutr. 2010 Dec;92(6):1522-7. doi: 10.3945/ajcn.2010.30185. Epub 2010 Oct 20. PMID 20962157
- [Derived] Ventura E, Davis J, Byrd-Williams C, Alexander K, McClain A, Lane CJ, Spruijt-Metz D, Weigensberg M, Goran M. Reduction in risk factors for type 2 diabetes mellitus in response to a low-sugar, high-fiber dietary intervention in overweight Latino adolescents. Arch Pediatr Adolesc Med. 2009 Apr;163(4):320-7. doi: 10.1001/archpediatrics.2009.11. PMID 19349560